CLINICAL TRIAL: NCT04799223
Title: Personalized Modulation of the Microbiota Through the Intelligent Design of Foods and Ingredients Based on Enterotype-Based Diagnosis (NUTRIBIOTA). Nutritional Intervention in Humans
Brief Title: Personalized Modulation of Microbiota
Acronym: NUTRIBIOTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Fermín Milagro Yoldi, Principal Investigator, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUTRIBIOTA
Record Dates: First submitted 2021-03-04; First posted 2021-03-16 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Microbial Colonization; Nutrition Disorders
Keywords: Obesity; Fecal microbiota; Nutrition; Diet; Insulin
MeSH Terms: conditions — Obesity; Communicable Diseases; Nutrition Disorders; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving the 4 designed foods (Experimental): The experimental group consumes the 4 foods designed for the study and will follow healthy eating guidelines.
  Interventions: Other: Four-foods eating guidelines
- Group with no designed foods (Active Comparator): The control group follows healthy eating guidelines.
  Interventions: Other: No designed-foods eating guidelines

INTERVENTIONS:
Other: Four-foods eating guidelines — To follow a healthy eating pattern and consume four (4) foods designed for the study (extra virgin olive oil with olive leaf extract, chickpea dish with spinach, vegetable cream dish, and olive fiber) and to follow a healthy eating pattern.
  Arms: Group receiving the 4 designed foods
Other: No designed-foods eating guidelines — To follow a healthy eating pattern. Their diet is not accompanied by the four newly designed foods of the other group.
  Arms: Group with no designed foods

SUMMARY:
Intestinal flora or microbiota is the group of bacteria that live in the intestine, in a symbiotic relationship with the human body. It is estimated that human beings have around 2,000 different bacteria species. The gut microbiota plays a key in many of the body's functions. Hence, the analysis of the gut microbiome provides insight into the state of the microbiota as an indicator of overall health due to its metabolic, protective and nutritional functions. A balanced diet promotes the formation and maintenance of a well-structured microbiota, in which the different species of microorganisms cohabit in a balanced and controlled system.

The study is based on the hypothesis that the intake of certain plant-based foods rich in various active ingredients (especially non-digestible carbohydrates, certain types of fats and polyphenols) can modulate the microbiota and thus improve the health status of the human population.

Taking into account this background, the objective of this study is to assess the effect of the inclusion of functional foods and ingredients within a balanced diet on the composition of the microbiota and also on health parameters associated with metabolic disease.

DETAILED DESCRIPTION:
The 60 volunteers participating in the study who meet the inclusion criteria, will be randomly divided into two groups:

* Control group (nutritional promotion): volunteers will be provided with basic nutritional recommendations based on a Mediterranean diet.
* Experimental group (Nutribiota): volunteers will be instructed to follow a dietary strategy similar to the control group, but including the functional foods and ingredients developed by the companies with the aim to promote a balanced and specific diet associated with improvements in the composition of the microbiota and metabolic parameters of the volunteers.

The duration of the study are 8 weeks, during which 4 visits are scheduled:

* Recruitment: this visit will consist on an initial screening in which the volunteers will be informed about the characteristics of the study and will be receive the information sheet and the informed consent form to be signed by all those interested in participating in the study. Volunteers who meet the inclusion for the study will be asked to complete the Food Frequency Questionnaire and Physical Activity Questionnaire for the next visit (visit 1). In addition, each participant will be provided with a faecal microbiota sample collection kit which they will have to hand in with the corresponding sample at the next visit (visit 1).
* Clinical investigation day 1 (week 0):after a fasting period of at least 10 hours, the nursing staff will take a blood sample to analyze the biochemical parameters and metabolomic profile. Anthropometric measurements will be taken from each volunteer (weight, height, waist and hip circumference, and body composition analysis by bioimpedance) with the collaboration of a dietician. In addition, faecal sample and Food Frequency Questionnaire and Physical Activity Questionnaire will be collected. Volunteers randomly assigned to the experimental group will be given the dishes and functional ingredients designed by the companies, which they will have to incorporate into a balanced dietary pattern following the indications given by the dietician.
* Clinical investigation day 2 (week 4): In this visit, the adherence of the volunteers to the study will be monitored and the weight of the volunteers will be registered. In addition, all study volunteers will be given a faecal microbiota sample collection kit, which should be handed in with the corresponding sample at the final visit. Moreover, Food Frequency Questionnaire and Physical Activity Questionnaire will be given to each volunteer in order to be filled for the final visit. Volunteers who belong to the experimental group will be given dishes and functional ingredients.
* Clinical investigation day 3 (week 8): Faecal sample, Food Frequency Questionnaire and Physical Activity Questionnaire will be collected. The procedures in this visit will be the same as in visit 1, but dishes and functional ingredients will not be given to the volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes with ages between 20 and 65 years.
* Volunteers with a body mass index between 24.9 and 34.9 kg / m2.
* Volunteers with intestinal dysbiosis.
* Physical examination and normal vital signs or clinically irrelevant for the study.
* Subjects must be able to understand and be willing to sign the informed consent.

Exclusion Criteria:

* Volunteers who have taken antibiotics or corticosteroids one month before the start of the intervention or antihistamines 15 days before the start of the intervention.
* Volunteers who are taken gastric protectors chronically.
* Volunteers who present changes in their pharmacological treatment in the last 3 months before the start of the study.
* Volunteers with intestinal pathologies (ulcerative colitis, Crohn's disease, or similar).
* Volunteers suffering from Covid-19

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Change of fecal microbiota composition | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Measured by analyzing the variable regions V3-V4 of the prokaryotic 16S rRNA (ribosomal ribonucleic acid) gene sequences, which gives 460 bp amplicons in a two-round PCR protocol. The kit used will be the Nextera® XT DNA Index Kit, FC-131-1002 (Illumina, San Diego, CA, USA).
  In the first step, PCR is used to amplify a template out of a DNA fecal sample using specific primers from Illumina. Then, sequencing libraries are built with the MiSeq® Reagent Kit v3 (600 cycles) MS-102-3003 (Illumina). Finally, paired-end sequencing is performed on a MiSeq platform (Illumina) with a 600 cycles Miseq run.
  Fecal samples are self-collected by the volunteers' fecal samples using OMNIgene.GUT kits from DNA Genotek (Ottawa, ONT, Canada), according to the standard instructions provided by the company

SECONDARY OUTCOMES:
Change of glucose concentration | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Glucose concentration will be reported in mg/dl
Change of total cholesterol concentration | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Total cholesterol concentration will be reported in mg/dl
Change of LDL-cholesterol concentration | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  LDL-cholesterol concentration will be reported in mg/dl by Friedewald equation.
Change of HDL-cholesterol concentration | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  HDL-cholesterol concentration will be reported in mg/dl
Change of triglyceride concentration | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Triglyceride concentration will be reported in mg/dl
Change of aspartate aminotransaminase concentration | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Aspartate aminotransaminase concentration will be reported in mg/dl
Change of alanine aminotransferase concentration | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Alanine aminotransferase concentration will be reported in U/L
Change of insulin concentration | Clinical The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).day 1 and 3
  Insulin concentration will be reported in U/L
Change of body weight | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Body weight will be reported in kg
Change of body mass index | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Body weight will be reported in kg
Change of body fat mass percentage | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Body fat mass will be reported in percentage
Change of body lean mass | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Body lean mass will be reported in kg
Change of body water percentage | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Body water will be reported in percentage
Change of visceral fat level | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Visceral fat level will be reported
Change of physical activity | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Physical activity level will be monitored by physical activity questionnaire
Change of dietary intake | The Time Frame contains two time points: day 1 (at baseline) compared to day 3 (after 8 weeks of dietary intervention).
  Dietary energy and macronutrient intake will be monitored by a food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fermín Milagro Yoldi, PhD, Principal Investigator — University of Navarra
Locations (1):
- Center for Nutrition Research. University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No